CLINICAL TRIAL: NCT03769584
Title: Follow-up of Treatment Outcome, Quality of Life, Sexual Life and Partnership After Surgery of Endometriosis
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-01728; sp18Tschudin
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Endometriosis
Keywords: quality of life; treatment outcome; sexuality; partnership; surgery of endometriosis
MeSH Terms: conditions — Endometriosis; Sexuality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Follow-up questionnaire — Online- Questionnaire investigating Follow-up of Treatment Outcome, Quality of Life, Sexual Life and Partnership After Surgery of Endometriosis
Other: Follow- up interview — Semi- structured Interview investigating Follow-up of Treatment Outcome, Quality of Life, Sexual Life and Partnership After Surgery of Endometriosis

SUMMARY:
Follow-up of treatment outcome, quality of life, sexual life and partnership after surgery of endometriosis by means of a questionnaire 1 year after surgical Intervention.

ELIGIBILITY:
Inclusion Criteria:

* surgery of endometriosis at Frauenklinik of University Hospital Basel (from 01.01.2017 until 31.12.2017)
* sufficient German language skills in order to be able to complete questionnaires

Exclusion Criteria:

* incapable of consenting

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with endometriosis undergoing surgery of endometriosis at Frauenklinik of University Hospital Basel (from 01.01.2017 until 31.12.2017)
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Endometriosis- associated symptoms assessed by questionnaire | 1 year after surgery of endometriosis
  questionnaire asking for pain (with menstruation, with sexual intercourse, with defecation, with urination) on a Visual Analogue Scale (VAS), ranging from 0 = no pain to 10 = intolerable pain
Treatment outcome of surgery of endometriosis assessed by VAS questionnaire | 1 year after surgery of endometriosis
  questionnaire asking for satisfaction with treatment outcome on a Visual Analogue Scale (VAS), ranging from 0 = absolutely dissatisfied to 10 = absolutely satisfied
Change in Quality of life assessed by questionnaire | before surgery of endometriosis and 1 year after surgery of endometriosis
  questionnaire asking for Quality of life on a Visual Analogue Scale (VAS), ranging from 0 = very bad to 10 = very good
Change in sexual life assessed by questionnaire | before surgery of endometriosis and 1 year after surgery of endometriosis
  questionnaire asking for Sexual life on a Visual Analogue Scale (VAS), ranging from 0 = absolutely dissatisfied to 10 = absolutely satisfied
Change in conduct of life assessed by questionnaire | before surgery of endometriosis and 1 year after surgery of endometriosis
  questionnaire asking for change in conduct of life (partnership, family, professional life, leisure activity, sportive activities) on a 6- item scale (ranging from "negative" to "positive")
Change in wish for child assessed by questionnaire | before surgery of endometriosis and 1 year after surgery of endometriosis
  questionnaire asking for change in wish for child on a 3- item scale (ranging from "yes" , "no answer" to "no")

SECONDARY OUTCOMES:
Follow-up of Treatment outcome of surgery of endometriosis assessed by interview | 1 year after surgery of endometriosis
  semi- structured interview to assess comments of study participants that are not depicted in the questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Sibil Tschudin, PD Dr. med, Principal Investigator — Frauenklinik Universitätsspital Basel
Locations (1):
- Frauenklinik University Hospital Basel, Basel, Switzerland